CLINICAL TRIAL: NCT06167876
Title: Safety and Efficacy of Stereotactic Body Radiotherapy in the Treatment of Hypertrophic Obstructive Cardiomyopathy: A Multicenter, Randomized, Single-blind, Controlled Study
Brief Title: Safety and Efficacy of Stereotactic Body Radiotherapy in the Treatment of Hypertrophic Obstructive Cardiomyopathy
Acronym: SAFECARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Shenghua Zhou, Professor, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LYG20230056
Record Dates: First submitted 2023-12-03; First posted 2023-12-13 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Hypertrophic Obstructive Cardiomyopathy; Stereotactic Body Radiotherapy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Radiosurgery; Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stereotactic Body Radiotherapy (SBRT) Treatment Group (Experimental): This arm of the study encompasses patients who are receiving the non-invasive Stereotactic Body Radiotherapy (SBRT) as the primary treatment for Hypertrophic Obstructive Cardiomyopathy (HOCM). The group will undergo precise imaging-guided radiotherapy targeting the interventricular septum, avoiding critical cardiac structures, and delivering a single high-dose radiation treatment with the aim of alleviating the symptoms of HOCM and improving cardiac function.
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT) Treatment
- Sham Procedure Control Group (Sham Comparator): Participants in this arm will undergo a sham procedure, which mimics the SBRT treatment process without actual radiation delivery. This group serves as a control to assess the efficacy and safety of the SBRT treatment by providing a comparative baseline. The sham procedure involves aligning patients with the linear accelerator and replicating the treatment environment, including equipment sounds and lighting, without administering any radiation.
  Interventions: Other: Sham Procedure

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy (SBRT) Treatment — The intervention in this study utilizes Stereotactic Body Radiotherapy (SBRT) for treating Hypertrophic Obstructive Cardiomyopathy (HOCM). The process begins with precise localization and planning, employing CT scans, Cardiac MRI (CMR), and echocardiography to accurately identify the target area in the interventricular septum, while avoiding critical structures like the aortic valve, His bundle, and left ventricular papillary muscles. Pre-treatment preparation involves using customized fixation devices to limit patient movement and breathing, coupled with cone-beam CT scans for accurate alignment with the Treatment Planning System (TPS). The treatment itself is delivered using image-guided linear accelerators, administering a single, focused dose of 25 Gy to the targeted area. This approach ensures precise radiation delivery, maximizing treatment efficacy while minimizing risks to surrounding cardiac tissues.
  Arms: Stereotactic Body Radiotherapy (SBRT) Treatment Group
Other: Sham Procedure — The sham procedure in this study is designed to closely mimic the actual Stereotactic Body Radiotherapy (SBRT) process without delivering any radiation. Participants in this arm are subjected to the same initial steps as those in the SBRT group, including precise alignment with the linear accelerator using CT scans and the application of customized fixation devices to limit movement and breathing. However, in this sham intervention, the linear accelerator is activated but does not emit any radiation. The procedure replicates the environmental aspects of the actual treatment, such as the equipment's sounds and lighting, to maintain the study's single-blind nature. This method ensures that participants in the sham group experience a procedure identical in appearance and feel to the SBRT treatment, without receiving any therapeutic dose, thereby serving as an effective control for evaluating the true impact of SBRT in treating HOCM.
  Arms: Sham Procedure Control Group

SUMMARY:
This study is designed to rigorously evaluate the safety and effectiveness of Stereotactic Body Radiotherapy (SBRT) as an innovative, non-invasive treatment for Hypertrophic Obstructive Cardiomyopathy (HOCM). HOCM, a prevalent cardiac condition, is primarily characterized by asymmetric septal hypertrophy, which results in the obstruction of the left ventricular outflow tract. This obstruction significantly compromises patient quality of life and is associated with severe risks, including arrhythmias and sudden cardiac death. While current treatments like medications, surgical septal myectomy, and percutaneous transluminal septal myocardial ablation (PTSMA) have proven to be effective, they are not without limitations. SBRT, a recent development in non-invasive cardiac radioablation, has shown encouraging results in early-stage studies, suggesting its potential as a safe and feasible option for HOCM treatment.

In this study, participants will be randomly assigned to either the SBRT treatment group or a control group receiving a sham procedure. The primary objective is to measure the change in the left ventricular outflow tract pressure gradient under provoked conditions, using cardiac ultrasound at a 6-month follow-up. This will provide a clear assessment of the direct impact of SBRT on the primary physiological complication of HOCM.

The study also sets forth several secondary objectives to provide a holistic view of the treatment's impact. These include evaluating changes in NYHA functional classification and KCCQ scores to assess improvements in symptom severity and quality of life, respectively. Additionally, we will monitor physical capacity through the 6-minute walk test, and biomarkers like NT-proBNP and cTNT for cardiac stress and damage. The effect of SBRT on QRS duration will be analyzed to understand its impact on cardiac electrical activity. The incidence of major adverse cardiac events (MACEs) within 6 months post-treatment will be recorded to evaluate safety, and the need for invasive septal reduction therapy post-treatment will be assessed to gauge long-term efficacy.

This study aims to provide a comprehensive understanding of the potential of SBRT as a treatment alternative for HOCM. By comparing its outcomes with those of traditional therapies, the study seeks to establish SBRT's role in symptom alleviation, quality of life enhancement, and risk reduction in HOCM management.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Confirmed diagnosis of Hypertrophic Obstructive Cardiomyopathy (HOCM) with a left ventricular outflow tract resting pressure gradient of 50mmHg or greater, as evidenced by cardiac ultrasound or Cardiac MRI.
* Willingness and consent to undergo non-invasive cardiac radioablation technology for the treatment of HOCM.
* Provision of informed consent, indicating voluntary participation in the study.
* Capability to read, understand, and communicate in Chinese for study-related procedures and consent.

Exclusion Criteria:

* Participation in any interventional clinical trial within 30 days prior to enrollment in this study, excluding participation in non-interventional and diagnostic reagent studies.
* Previous receipt of any invasive treatment options for HOCM.
* Advanced heart failure characterized by NYHA functional class IV.
* A left Ventricular Ejection Fraction (LVEF) of less than 30%.
* Concurrent severe illnesses that are life-limiting with an expected lifespan of less than one year.
* Planned or requirement for any form of surgical intervention.
* Pregnancy or currently breastfeeding.
* Involvement in the execution or implementation of this study, including study staff and their immediate family members.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Change in Left Ventricular Outflow Tract Pressure Gradient under Provoked Conditions | 6 months post-treatment
  This primary outcome measure evaluates the effectiveness of non-invasive radiotherapy (SBRT) in altering the left ventricular outflow tract pressure gradient under provoked conditions in patients with Hypertrophic Obstructive Cardiomyopathy (HOCM). The measurement is determined using cardiac ultrasound, assessing the extent to which SBRT can alleviate the obstruction in the heart's outflow tract, a key indicator of therapeutic success in HOCM treatment.

SECONDARY OUTCOMES:
Change in Left Ventricular Outflow Tract Pressure Gradient under Resting Conditions | 6 months post-treatment
  This measure assesses the change in the left ventricular outflow tract pressure gradient under resting conditions in HOCM patients, using cardiac ultrasound at a 6-month follow-up. It aims to evaluate the impact of non-invasive SBRT treatment on cardiac function during periods of rest.
Impact on NYHA Functional Classification | 6 months post-treatment
  This outcome evaluates the effect of SBRT on the NYHA functional classification of patients, indicating changes in symptomatic heart failure and overall cardiac performance post-treatment.
Changes in Kansas City Cardiomyopathy Questionnaire (KCCQ) Scores | 6 months post-treatment
  This measure evaluates the effect of treatment on patient quality of life and symptomatic relief. It is quantified using the Kansas City Cardiomyopathy Questionnaire (KCCQ), a comprehensive scale that measures heart failure symptoms and their influence on daily activities. The KCCQ scale ranges from 0 to 100, where higher scores indicate better health status and lower scores signify worse outcomes. This scale effectively captures the patient's experience and the impact of heart failure on their quality of life.
Performance in the 6-Minute Walk Test | 6 months post-treatment
  This outcome evaluates the physical capacity of patients post-treatment, measured through the 6-minute walk test, a standard test of aerobic capacity and endurance.
Concentration Changes of NT-proBNP and cTNT Post-SBRT Treatment | 6 months post-treatment
  This measure monitors the levels of NT-proBNP and cTNT, biomarkers of cardiac stress and damage, post-SBRT treatment, providing insights into the physiological changes within the heart.
Impact on QRS Duration | 6 months post-treatment
  This outcome analyzes the effect of SBRT on QRS duration, assessed through electrocardiogram (ECG), to understand any changes in cardiac electrical activity post-treatment.
Incidence of Major Adverse Cardiac Events (MACEs) | 6 months post-treatment
  This measure tracks the occurrence of major adverse cardiac events within 6 months post-treatment, offering crucial data on the safety profile of SBRT in treating HOCM.
Monitoring of Serious Adverse Events (SAEs) | Up to 6 months post-treatment
  This measure involves meticulous monitoring of any serious adverse events during and after treatment, ensuring a comprehensive safety assessment of SBRT as a therapeutic approach.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Hunan Provincial People's Hospital, The First Affiliated Hospital of Hunan Normal University, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of University of South China, Hengyang, Hunan
  - Xiangtan Central Hospital, Xiangtan, Hunan

IPD SHARING:
Plan to Share IPD: No